CLINICAL TRIAL: NCT06496269
Title: Impact of Microvascular Inflammation on Kidney Allograft Outcome: a Multinational Cohort Study
Brief Title: Impact of Microvascular Inflammation on Kidney Allograft Outcome
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: MVI_Kidney_002
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Transplant;Failure,Kidney; Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Graft microvascular inflammation poses a significant challenge to successful kidney transplantation due to its heterogeneous clinical presentation. There is a critical need to unravel the clinical significance of newly defined allograft microvascular inflammation phenotypes in the Banff 2022 classification and assess the implications of these new phenotypes on kidney transplant precision diagnostics and patient risk stratification.

DETAILED DESCRIPTION:
Antibody-mediated rejection is a major cause of graft failure in kidney transplant recipients, with allograft microvascular inflammation serving as the hallmark histological lesion of antibody-mediated graft injury. However, the frequent occurrence of graft microvascular inflammation in the absence of circulating anti-HLA donor-specific antibodies highlights the incomplete understanding of the mechanisms underlying this inflammation. This heterogenous presentation poses a significant challenge in the clinical setting, as current treatment strategies often prove ineffective, hindering the improvement of allograft and patient care. The Banff 2022 classification update has reappraised lesions of microvascular inflammation, identifying new diagnostic phenotypes of microvascular inflammation. However, the clinical significance of these phenotypes is yet to be determined.

The aims of this study are:

1. To determine the impact of the revised Banff 2022 Classification on the diagnostic classification of phenotypes related to microvascular inflammation, compared to previous Banff 2019 Classification.
2. To assess the association of microvascular inflammation phenotypes with kidney allograft survival.
3. To assess the association of microvascular inflammation phenotypes with disease progression, defined by transplant glomerulopathy occurrence (cg and subsequent antibody-mediated rejection episodes.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients, with at least one kidney transplant biopsy performed, assessed with the Banff classification.

Exclusion Criteria:

* Missing data for a rejection-related diagnosis according to the 2019 and 2022 Banff classification.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients of all sexes recruited in observational studies performed in Europe and United States, with at least one kidney biopsy performed with all the relevant data to provide a diagnosis according to the 2019 and 2022 Banff classification, including clinical data (recipient and donor's age, sex and transplant characteristics).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Microvascular inflammation-related diagnoses according to the Banff 2022 Classification | March 2004 to December 2023
Kidney allograft loss | March 2004 to December 2023

SECONDARY OUTCOMES:
Transplant glomerulopathy | March 2004 to December 2023
(Recurrent) antibody-mediated rejection episode | March 2004 to December 2023

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Principal Investigator — Paris Institute for Transplantation and Organ Regeneration
Locations (19):
- United States (7):
  - Pediatric Nephrology, UCLA Mattel Children's Hospital, Los Angeles, California
  - Division of Pediatric Nephrology, Children's Pediatric Institute, Atlanta, Georgia
  - Division of Pediatric Nephrology, Children's Mercy Hospital, Kansas City, Missouri
  - Acute Dialysis Units, Pediatric Kidney Transplant, Charleston, South Carolina
  - Division of Pediatric Nephrology and Hypertension, Le Bonheur Children's Hospital, Memphis, Tennessee
  - Department of Pediatrics, Seattle Children's Hospital, Seattle, Washington
  - Division of Nephrology, Department of Medicine, University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- France (9):
  - Bordeaux University Hospital, Department of Nephrology, Transplantation, Dialysis and Apheresis, Bordeaux
  - Department of Transplantation, Nephrology and Clinical Immunology, Hospices Civils de Lyon, Lyon
  - Department of Nephrology, Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Nantes University Hospital, Department of Nephrology, Nantes
  - Division of Pediatric Nephrology, Necker Hospital, AP-HP, Paris
  - Division of Pediatric Nephrology, Robert Debré Hospital, AP-HP, Paris
  - Kidney Transplant Department, Necker Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Kidney Transplant Department, Saint-Louis Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Department of Nephrology-Dialysis-Transplantation, Centre Hospitalier Universitaire de Toulouse, Toulouse
- Department of Nephrology and Critical Care Medicine, Charité - Universitätsmedizin Berlin, Freie Universität Berlin, Berlin Institute of Health, Berlin, Germany
- Department of Nephrology and Kidney Transplantation, Vall d'Hebrón University Hospital, Barcelona, Spain
- Division of Abdominal and Transplantation Surgery, Department of Surgery, Geneva University Hospitals,, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The data analyzed during the current study are available on reasonable request including standards for General Data Protection Regulation and Institutional Review Board approval.

REFERENCES:
- [Derived] Sablik M, Sannier A, Raynaud M, Goutaudier V, Divard G, Astor BC, Weng P, Smith J, Garro R, Warady BA, Zahr RS, Twombley K, Dharnidharka VR, Dandamudi RS, Fila M, Huang E, Sellier-Leclerc AL, Tonshoff B, Rabant M, Verine J, Del Bello A, Berney T, Boyer O, Catar RA, Danger R, Giral M, Yoo D, Girardin FR, Alsadi A, Gourraud PA, Morelon E, Le Quintrec M, Try M, Villard J, Zhong W, Bestard O, Budde K, Chauveau B, Couzi L, Brouard S, Hogan J, Legendre C, Anglicheau D, Aubert O, Kamar N, Lefaucheur C, Loupy A. Microvascular Inflammation of Kidney Allografts and Clinical Outcomes. N Engl J Med. 2025 Feb 20;392(8):763-776. doi: 10.1056/NEJMoa2408835. Epub 2024 Oct 24. PMID 39450752